CLINICAL TRIAL: NCT05118269
Title: Targeted Segmental Vapor Ablation Treatment of Emphysema With Upper Lobe Predominance: A Randomized Controlled Trial of InterVapor® in France - The TARGET Trial
Brief Title: A Randomized Controlled Trial of InterVapor® in France - The TARGET Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor made the decision not to conduct this study. No subjects were treated in the study and all centers closed.
Sponsor: Uptake Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-2250
Record Dates: First submitted 2020-07-08; First posted 2021-11-11 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Emphysema
Keywords: Heterogeneous; Thermal Vapor; Ablation; Bronchoscopy; LVR; Lung Volume Reduction
MeSH Terms: conditions — Emphysema | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio between treatment group and control group. Subjects randomized to the Control Group may be allowed to cross over to the treatment group and offered the InterVapor treatment at 12 months, once they have completed the protocol defined follow-up period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment plus Optimal Medical Therapy (Experimental): Patients will be treated with the InterVapor System and Optimal Medical Therapy
  Interventions: Device: Treatment plus Optimal Medical Therapy
- Optimal Medical Therapy (Control) (Active Comparator): Patients will be treated according to Optimal Medical Therapy
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Device: Treatment plus Optimal Medical Therapy — Patients will be treated with the InterVapor System in 1 to 2 segments in the upper lobes of each lung (2 to 3 segments total). Patients will also receive Optimal Medical Therapy. Guidelines for prescribing medical treatment for emphysema are published by the American Thoracic Society (ATS) and the National Heart Lung and Blood Institute/World Health Organization (NHLBI/World Health Organization , Global Initiative for Chronic Obstructive Lung Disease (GOLD) workshop summary).
  Other Names: InterVapor; BTVA
  Arms: Treatment plus Optimal Medical Therapy
Other: Optimal Medical Therapy — Patients will receive Optimal Medical Therapy. Guidelines for prescribing medical treatment for emphysema are published by the American Thoracic Society (ATS) and the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO GOLD workshop summary).
  Arms: Optimal Medical Therapy (Control)

SUMMARY:
This study is designed to prospectively document changes in FEV1 and health-related quality of life 12 months following sequential segmental treatment with InterVapor® in patients with heterogeneous emphysema with upper lobe predominance. For validity of the study, the results will be compared to patients that receive optimal medical therapy.

DETAILED DESCRIPTION:
The primary objectives are to prospectively document changes in FEV1 and health-related quality of life 12 months following sequential segmental treatment with Bronchoscopic Thermal Vapor Ablation (BTVA) using the InterVapor system in patients with heterogeneous emphysema with upper lobe predominance. The French TARGET trial is a prospective, multi-center, single blind, randomized controlled study. 150 participants will be enrolled in the study (1:1 randomization with 75 InterVapor, 75 controls) with a 24-month follow-up period. Subjects randomized to the Control Group may be allowed to cross over to the treatment group and offered the InterVapor treatment once they have completed the protocol defined 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and ≤ 80 years old
2. Heterogeneous emphysema with upper lobe predominance in at least one lung segment to be treated (defined as a Heterogeneity Index (HI) ≥ 1.2 per CT)
3. Post-bronchodilator FEV1 ≥ 15% and ≤ 45% of predicted value
4. Total lung capacity (TLC) ≥ 100% predicted
5. Post-bronchodilator Residual volume (RV) ≥ 200% predicted
6. 6-minute walk distance (6MWD) > 100m and ≤ 450m
7. (Partial Pressure of Oxygen) PaCO2 ≤ 45 mm Hg; PaO2 > 45 mm Hg on room air
8. Non-smoking for 4 months prior to study enrollment as confirmed by:

   1. negative urine analysis or serum cotinine level of ≤ 10 ng/mL, or negative CO Hb test OR
   2. If using smoking cessation product(s) containing nicotine at screening, serum cotinine level ≤ 13.7 ng/ml (or arterial carboxyhemoglobin ≤ 2.5%)
9. Optimized medical management (consistent with GOLD guidelines)

   1. Pharmacological:

1.Long acting bronchodilator (LABA),Long-acting muscarinic antagonists (LAMA), LAMA + LABA, or LABA + ICS > 1 year

b. Evidence of completed Pulmonary Rehabilitation

1. ≥ 6 weeks out-patient or ≥ 3 weeks in-patient within 12 months of enrollment; or,
2. Patient has or continues to participate in at home rehabilitation program (i.e. a walking program) within 6 weeks of enrollment under the supervision of a health care professional

10. Mentally and physically able to provide written informed consent to participate in the study. Protected people as defined by the Code de la Sante Publique cannot be included in the study

Exclusion Criteria:

1. DLCO < 20% predicted
2. Uncontrolled pulmonary hypertension (systolic pulmonary arterial pressure >45 mm Hg) or evidence or history of cor pulmonale as determined by recent echocardiogram
3. Clinically significant bronchiectasis
4. Clinically significant (greater than 4 tablespoons per day) sputum production.
5. Two (2) or more COPD exacerbations or pneumonia episodes requiring hospitalization in the last year
6. Evidence of active infection in the lungs at the time of procedure.
7. Daily use of systemic steroids, > 10 mg prednisolone (or equivalent) daily.
8. Lung pathology of nodule not proven stable or benign
9. Clinically significant pulmonary fibrosis
10. Prior lung transplant, lung volume reduction surgery (LVRS), bullectomy, or lobectomy
11. Prior lung volume reduction via endobronchial valves(s), coil(s), and/or polymer. Note: Patients whose endobronchial valves have been removed can be treated if: all valves removed ≥ 3 months prior to InterVapor and baseline bronchoscopy reveals no airway obstruction or obvious tissue granulation
12. Large bulla (defined as > 1/3 volume of the lobe)
13. Highly diseased upper and lower lobes in contralateral lung (%-950 HU density >50%)
14. Paraseptal emphysema in any segment targeted for treatment
15. Myocardial Infarction or congestive heart failure within 6 months of screening.
16. Diagnosis of heart failure with Left Ventricular Ejection Fraction (LVEF) < 45% as determined by recent echocardiogram (completed within 3 months prior to screening).
17. Unable to safely discontinue anti-coagulants or platelet inhibitors for 6 weeks post procedure.
18. Body mass index (BMI) > 32 kg/m2
19. Patient taking immunosuppressive drugs for the treatment of cancer, rheumatic arthritis, autoimmune disease, or prevention of tissue or organ rejection.
20. Subject is pregnant or lactating, or plan to become pregnant within the study timeframe
21. Any disease or condition that is likely to limit survival to less than one year
22. Concomitant illnesses or medications that may pose a significant increased risk for complications following treatment with InterVapor®
23. Currently enrolled in another clinical trial studying an experimental treatment.
24. Any condition that would interfere with completion of the study including study assessments and study procedure including bronchoscopy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Changes in FEV1 between Treatment vs Control at 12 months | 12 months
  Percentage change in Forced expiratory volume in 1 second (FEV1) compared to active comparator: Change in FEV1, percent change from baseline to 12 months in FEV1, where FEV1 is expressed in raw units of volume (mL).
St. George's Respiratory Questionnaire for patients with Chronic Obstructive Pulmonary Disease (SGRQ-C) changes between Treatment vs Control at 12 months | 12 months
  Health-related Qualify of Life (SGRQ-C) compared to active comparator. This is calculated as change from baseline to 12 months in SGRQ-C Total Score. SGRQ-C scores range from 0 to 100. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Improvement in other measures of pulmonary function- Forced Expiratory Volume, absolute change- at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Change in FEV1, abs: Absolute change from baseline to follow-up in FEV1, where FEV1 is expressed in raw units of volume (mL).
Improvement in other measures of pulmonary function- Forced Expiratory Volume, Percent change- at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Change in FEV1, Percent Predicted value: Percent change from baseline to follow-up in FEV1, where FEV1 is expressed in percent predicted computed by European Respiratory Standard (ERS) standards.
Improvement in other measures of pulmonary function- Forced Expiratory Volume, Abs, PP change- at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Change in FEV1, abs, PP: absolute change from baseline to follow-up in FEV1, where FEV1 is expressed in percent predicted computed by ERS standards.
Improvement in other measures of pulmonary function- Forced Vital Capacity(FVC) change- at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Change in FVC: percent change from baseline to follow-up in Forced Vital Capacity, expressed in raw units of volume(mL)
Improvement in other measures of pulmonary function- Forced Vital Capacity Percent Predicted change- at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Change in FVC PP: percent change from baseline to follow-up in Forced Vital Capacity, expressed in percent predicted computed by ERS standards
Improvement in other measures of pulmonary function- Residual Volume- at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Percent change from baseline to follow-up in Residual Volume
Improvement in other measures of pulmonary function- Residual Volume-Abs at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Percent change from baseline to follow-up in Residual Volume, where RV is expressed in raw units of volume (mL).
Improvement in other measures of pulmonary function- Residual Volume-Percent Predicted value at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Percent change from baseline to follow-up in Residual Volume, where RV is expressed in percent predicted computed by ERS standards.
Improvement in other measures of pulmonary function- Residual Volume-Abs Percent Predicted value at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Absolute change from baseline to follow-up in Residual Volume, where RV is expressed in percent predicted computed by ERS standards
Improvement in other measures of pulmonary function-Diffusing Capacity of Lung (DLCO)- Percent Predicted Value at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Percent change from baseline to follow-up in Diffusing Capacity of the Lungs for Carbon Monoxide, where DLCO is expressed in percent predicted computed by ERS standards.
Improvement in other measures of pulmonary function-Diffusing Capacity of Lung (DLCO)- Absolute Percent Predicted Value at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Absolute change from baseline to follow-up in Diffusing Capacity of the Lungs for Carbon Monoxide, where DLCO is expressed in percent predicted computed by ERS standards.
Changes in segmental lung volumes from as assessed by CT at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Changes in segmental lung volumes from baseline to 12 months as assessed by CT
Changes in pulmonary function tests as assessed by body plethysmography measures at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Changes in pulmonary function tests as assessed by body plethysmography measures at 12 months
Number of serious adverse events and fatal events | 12 months, 18 months, 24 months
  Number of serious adverse events (SAEs) and fatal events
Binary responder analysis to determine minimally clinical important difference for FEV1 at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Binary responder analysis to determine Minimal Clinically Important Difference (MCID) for the following:
  • FEV1 (> 12% predicted) in Treatment vs Control at 12 months
Binary responder analysis to determine minimally clinical important difference for SGRQ-C at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Binary responder analysis to determine Minimal Clinically Important Difference (MCID) for the following:
  • SGRQ (> 8 points) in Treatment vs Control at 12 months
Binary responder analysis to determine minimally clinical important difference for 6 Minute Walk Distance (6MWD) at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Binary responder analysis to determine Minimal Clinically Important Difference (MCID) for the following:
  • 6MWD (> 26m) in Treatment vs Control at 12 months
Binary responder analysis to determine minimally clinical important difference for COPD Assessment Test (CAT) score at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Binary responder analysis to determine Minimal Clinically Important Difference (MCID) for the following:
  • CAT Score (> 2 points) in Treatment vs Control at 12 months
Binary responder analysis to determine minimally clinical important difference for Shortness of Breath Questionnaire (SOBQ) score at 12, 18 and 24 months | 12 months, 18 months, 24 months
  Binary responder analysis to determine Minimal Clinically Important Difference (MCID) for the following:
  • SOBQ Score (> 5 points) in Treatment vs Control at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guibert, Prof, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Centre Hospitalier Universitaire de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No